CLINICAL TRIAL: NCT02326545
Title: MindLight: A Video Game Intervention to Reduce Children's Anxiety
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Dr. Tom Hollenstein, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MindLight
Record Dates: First submitted 2014-12-15; First posted 2014-12-29 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Anxiety
Keywords: Video Games; Child; Adolescent
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MindLight (Experimental): MindLight is the video game being tested for effectiveness to reduce child anxiety
  Interventions: Behavioral: MindLight
- Online CBT (Active Comparator): Online CBT program for children
  Interventions: Behavioral: Online CBT

INTERVENTIONS:
Behavioral: MindLight — MindLight is a video game that uses neurofeedback as part of game mechanics. Participants play for 5 hours total over 3 weeks. Measures taken pre, post, and 3-month follow-up.
  Arms: MindLight
Behavioral: Online CBT — Five sessions of power point slides that cover primary concepts and homework of cognitive behavioral therapy. Adapted for children. Measures taken pre, post, and 3-month follow-up.
  Other Names: Cognitive Behavioral Therapy
  Arms: Online CBT

SUMMARY:
Anxiety is the most prevalent form of children's mental health problems and demand far exceeds treatment availability. Even when children do have access to care, evidence-based treatments such as cognitive-behavioural therapy have several limitations: they are largely didactic, leaving children unmotivated and disengaged; children get little practice in using the skills they are taught, creating a large gap between their knowledge and their everyday behaviour and therapy is costly, often prohibitive for the children that most need it. Therapeutic video games can address each of these gaps: they are engaging contexts through which children practice skills (rather than memorize lessons), and they cost substantially less than conventional approaches. The proposed research will test the effectiveness of MindLight, an innovative video game that targets childhood anxiety problems. MindLight incorporates several evidence-based strategies including relaxation and exposure techniques, attention bias modification methods, and neurofeedback mechanics that together produce an immersive game world through which children learn to manage and overcome anxiety symptoms. Two randomized controlled studies with 8-16 year old children are proposed to test the effectiveness of MindLight in reducing anxiety: the first is a prevention study aimed at children at risk for developing serious anxiety problems and the second is a clinical trial aimed at decreasing symptoms in anxiety-disordered children. Children randomly assigned to the intervention group will play MindLight for 5 hours over 2-3 weeks; control participants in the prevention sample will play a commercial video game with a similar theme for the same amount of time whereas control participants in the clinical sample will use an online cognitive behavioural therapy (CBT) program. Both studies will assess children's anxiety levels before the intervention, just after, and at a 3-month follow-up. Moderators (e.g., comorbidities) and mediators (e.g., attention biases) will be assessed to identify potential mechanisms of change associated with successful intervention effects.

DETAILED DESCRIPTION:
Over the next two years, the investigators will be collecting data on two samples, henceforth identified as the Clinical Sample and Prevention Sample. The laboratory protocol (pre, post, and follow-up) is the same for each; however the screening and recruitment are not. In this section, only those procedures and methods of the lab visit that are common to both are described. Next the video game intervention procedures are described. Participant and recruitment details are in subsequent sections.

Each participant will visit the Adolescent Dynamics Lab three times (pre, post, and follow-up) with only minor differences where noted. Parents will accompany children to the lab and, following the completion of consent forms (pre only), complete a set of questionnaires via computer:

Child report:

* Demographics
* Spence Child Anxiety Scale (SCAS)
* Strengths and Difficulties Questionnaire (SDQ)- emotional symptoms
* Top Problems questionnaire (TP)
* Coping Questionnaire
* Self-Efficacy Questionnaire (SEQ-C)

Parent report:

* Demographics (including what interventions for child's mental health have been tried)
* SCAS (report on child)
* Strengths and Difficulties Questionnaire - emotional symptoms (report on child)
* Depression, Anxiety and Stress Scale-21 (DASS21, report on self)

Questionnaires at Post are the same as Pre and Follow-up except for addition of Video game evaluation (child report).

Once questionnaires are completed, the child participant will have sensors for psychophysiological recording attached by a female experimenter. First, two sensors for recording electrodermal response (aka galvanic skin response or skin conductance) will be attached to the tips of the second and third finger of the non-dominant hand. Children's fingers will be wiped clean before applying a dab of conducting gel on the two fingers and affixing the sensors with Velcro straps firmly but not uncomfortably. Next, two sticker electrodes for measuring electrocardiogram signals (e.g., heart rate) are applied in a Lead-II configuration: one affixed just below the right collarbone and the other on the side of the torso near the lower left rib. These circular stickers (about the size of a Loonie) have a metal nub to which wires are affixed via clips. Finally, a respiration belt is wrapped around the torso below the breast or pectoral muscle outside of the clothing. The belt is elastic and registers the expansion and contraction due to respiration. All three measurement devices are attached to a Biopac TEL-100 battery pack attached to the back of the participant's chair. This device is then attached to a computer in the adjacent room via the Biopac MP-150 amplifier. Physiological signals are recorded using AcqKnowledge 4.2 software from Biopac. The child and parent will be able to observe the signals as they will be recorded via a monitor in the observation room.

Once the sensors and physiological recording has been set up, the parent will be asked to leave the room and wait in a room nearby until the child has completed the tasks. The sequence of tasks is:

1. Baseline Physiology (3 tasks): (a) equipment baseline: watch a neutral film to allow the measurements to settle(2 minutes), (b) paced breathing to get resting respiratory sinus arrhythmia (RSA; a measure of parasympathetic activity) while participants breathe in and out in synch with a bar that goes up and down at 9 cycles per minute displayed on a monitor (2 minutes), and (c) pre-task baseline for calculating reactivity to social and cognitive stress (2 minutes)
2. Attention bias task: dot probe task. (5 minutes)
3. Social Stress Task: spontaneous speech on any topic of the child's choosing (3 minutes).
4. Quick self-report of feelings (< 1 minute)
5. Recovery 1: participant sits alone in the observation room quietly to assess return to baseline levels of arousal (3 minutes).
6. Cognitive Stress Task: counting backwards by 7's from 2148. Incorrect answers will require the participant to start over from the beginning (2 minutes)
7. Recovery 2: participant sits alone in the observation room quietly to assess return to baseline levels of arousal (3 minutes).

Finally, the parent will be brought back into the room as the sensors are removed. Debriefing will occur only after the final follow-up lab visit. Anticipated time to complete lab visit is approximately one hour.

MINDLIGHT GAME PLAY Participants in the treatment condition will play 5 total hours of MindLight, one hour at each sitting, over the course of 2-3 weeks. Game play will occur either in schools or at the participant's home. For the Prevention Sample, MindLight will be played in participating middle and high schools in the Limestone District School Board. Participants in the Clinical Sample who attend these schools will also play the game at the school. However, for children recruited through the Hotel Dieu Mood and Anxiety clinic (see recruitment details) who do not attend one of the participating schools will play MindLight at home. In all cases, a research assistant will be present to set up the game and monitor any equipment difficulties.

To play the game, children will wear a lightweight MindWave headset that has a single electrode that must touch the forehead (see attached images). There is a clip that attaches comfortably to the earlobe as well. The electroencephalogram (EEG) signals in the alpha, beta, and gamma frequencies are used to extract two continuous signal streams that are measures of focused attention and arousal. These signals are used in the game to control the character's "mind light," a magical hat he wears that has a light on the end of a signal antenna, by focusing a beam of light toward specific targets to solve puzzles within the game and expanding the range of light inversely proportional to the degree of arousal. Thus, children control key aspects of the game with their mind.

Control participants in the Prevention Sample will play Max and the Magic Marker, a commercially available game with similar features to MindLight but without the key mechanisms targeting anxiety reduction (attention bias modification and relaxation). The amount of game play time and location will be the same as those in the intervention group.

ONLINE COGNITIVE BEHAVIOURAL THERAPY Control participants in the Clinical Sample will receive an online version of cognitive behavioural therapy (CBT) based on the skills taught in Mind over Mood by D. Greenberger and C. Padesky. The program provides general information on each topic, an overview on helpful skills, and homework sheets by email that directly corresponds with how a live, 8-week group therapy session would be conducted. Participants will also receive feedback on homework on a specific day every week from a therapist at Hotel Dieu.

Description of participants CLINICAL SAMPLE Children 8-16 years old who have made an appointment at the Mood and Anxiety Clinic at Hotel Dieu specifically for problems with anxiety. Only those with autism or significant developmental delays will be excluded. The investigators will recruit 100 children, with half randomly assigned to the MindLight intervention group.

PREVENTION SAMPLE Children 10-16 years old attending participating schools in the Limestone District School Board who have been identified as having elevated anxiety symptoms via a self-report measure of anxiety. Only those with autism or significant developmental delays will be excluded. The investigators will recruit 100 children, with half randomly assigned to the MindLight intervention group.

Recruitment details CLINICAL SAMPLE Participants will be recruited following initial assessment at the Hotel Dieu Mood and Anxiety Clinic. The typical wait period between this initial diagnostic assessment and the start of either group or one-on-one therapy is 3-6 months. Our intervention will occur during this wait period. During the initial assessment at the clinic, children aged 8-16 will be invited to participate in the study. They will be provided a brief explanation of the study and will indicate to the clinician whether they give permission to be contacted by the recruitment coordinator who will provide all of the details of the study. The participant will be made aware that they are under no obligation to participate in the study by agreeing to be contacted. Those who assent to participate will be invited to the Adolescent Dynamics Lab to begin participation.

PREVENTION SAMPLE Children in grades 6-10 who attend one of the participating schools will complete one questionnaire during class time, the Spence Children's Anxiety Scale (SCAS). Children who score 1 standard deviation above the mean for (a) the total score or (b) two of the subscales (not including the obsessive-compulsive scale) will be considered at risk for developing an anxiety disorder. These children will be invited to participate in the study by visiting the Adolescent Dynamics Lab. Consent for the study will be obtained from the parent prior to the SCAS screening.

ELIGIBILITY:
Inclusion Criteria:

* Elevated levels or clinical diagnosis of anxiety

Exclusion Criteria:

* Developmental disorders or autism

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in Spence Children's Anxiety Scale following intervention | Pre-Tx (1st lab visit), Post-Tx (2nd lab visit 3 weeks later), Follow-up (final lab visit 3 months later)
  Widely used scale for measuring children's anxiety will be used to determine the degree of reduction in anxiety symptoms immediately following the intervention and whether this reduction is maintained at a 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hollenstein, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared

REFERENCES:
- [Derived] Tsui TYL, DeFrance K, Khalid-Khan S, Granic I, Hollenstein T. Reductions of Anxiety Symptoms, State Anxiety, and Anxious Arousal in Youth Playing the Videogame MindLight Compared to Online Cognitive Behavioral Therapy. Games Health J. 2021 Oct;10(5):330-338. doi: 10.1089/g4h.2020.0083. Epub 2021 Aug 17. PMID 34403591